CLINICAL TRIAL: NCT00104559
Title: Interactive Multimedia Informed Consent (iMIC) for HIV Research
Brief Title: Computer-Generated Vs. Standard Informed Consent for HIV Research Studies
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Brian D. Raffety, PhD, The Circumplex Company
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 1R43AI058870-01 (NIH); 1R43AI058870-01 (NIH)
Record Dates: First submitted 2005-03-01; First posted 2005-03-02 (Estimated); Last update posted 2008-09-26 (Estimated); Status verified 2008-09

CONDITIONS: HIV Infections
Keywords: HIV; Informed Consent
MeSH Terms: conditions — HIV Infections

ARMS (4):
- 1 (Experimental): Participants will receive the computer-based tutorial for VT and then the standard paper consent form for AT
  Interventions: Behavioral: iMIC-generated consent form and tutorial; Behavioral: Standard paper consent form
- 2 (Experimental): Participants will receive the standard paper consent form for VT and then the computer-based tutorial for AT
  Interventions: Behavioral: iMIC-generated consent form and tutorial; Behavioral: Standard paper consent form
- 3 (Experimental): Participants will receive the computer-based tutorial for AT and then the standard paper consent form for VT
  Interventions: Behavioral: iMIC-generated consent form and tutorial; Behavioral: Standard paper consent form
- 4 (Experimental): Participants will receive the standard paper consent form for AT and then the computer-based tutorial for VT
  Interventions: Behavioral: iMIC-generated consent form and tutorial; Behavioral: Standard paper consent form

INTERVENTIONS:
Behavioral: iMIC-generated consent form and tutorial — Computer-based consent form and tutorial
Behavioral: Standard paper consent form — Standard paper consent form

SUMMARY:
The purpose of this study is to test an interactive multimedia informed consent (iMIC) computer program to see if the program can generate a consent form that potential participants in an HIV trial can understand. This study will also determine if these participants prefer the computer-generated consent form and associated interactive tools to a standard consent form written by researchers.

Study hypothesis: 1) Participants who receive information about clinical trials from iMIC Consent Tutorials will answer more questions about the trial correctly than participants who receive information about clinical trials from standard paper consent forms. 2) Participants will rate the iMIC Consent Tutorials as having better usability and user satisfaction than standard paper consent forms.

DETAILED DESCRIPTION:
Researchers conducting clinical trials have a legal and ethical obligation to provide participants key information about the trial so that they may either decline participation or grant their informed consent to participate in the study. However, information provided to prospective clinical trial participants is often complex and confusing; often, language used in informed consent is written far above participants' reading level. This study will evaluate the usefulness of a consent form authoring system that helps researchers write comprehensive and understandable consent forms; the authoring system produces both paper consent forms and interactive computer tutorials that are designed to teach potential volunteers about the research study they are considering. This study will compare iMIC-generated consent forms and computer tutorials with standard consent forms for two mock HIV studies: a vaccine trial (VT) and an antiretroviral drug trial (AT).

The iMIC software provides researchers a computer-based authoring environment for producing easier-to-understand informed consent documents. iMIC assists researchers by helping them focus on clearly defining consent issues and content goals, including regulatory, legal, and ethical guidelines to be followed. Through tests for readability and other feedback, iMIC ensures that all the content requirements of good informed consent are met. iMIC generates a paper consent form and an interactive multimedia computer tutorial to help volunteers learn about the clinical trial. The paper consent document can be stand alone or used in conjunction with the generated computer tutorial.

Each participant will receive two consent interventions: one computer-based tutorial and one standard paper consent form. Participants will be randomly assigned to one of four groups. Group 1 will receive the computer-based tutorial for VT and then the standard paper consent form for AT. Group 2 will receive the standard paper consent form for VT and then the computer-based tutorial for AT. Group 3 will receive the computer-based tutorial for AT and then the standard paper consent form for VT. Group 4 will receive the standard paper consent form for AT and then the computer-based tutorial for VT.

At the start of the session, participants will be asked demographic questions and will receive the first consent intervention. When they have completed the intervention, they will be asked 15 questions about the key elements of the clinical trial they have just learned about, as well as an additional series of usability and satisfaction questions about the consent intervention. Next, they will receive the second consent intervention that will teach them about the second clinical trial. Again, they will be asked knowledge and usability and satisfaction questions. After completing the second consent intervention, participants will be asked to compare and answer questions about the two methods of receiving information about clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected OR at risk for HIV infection
* Able to read English at the 5th grade level

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-01; Primary Completion 2007-07 (Estimated); Study Completion 2009-03 (Estimated)

PRIMARY OUTCOMES:
Clinical trial knowledge acquisition | Throughout study
Consent form usability | Throughout study
Volunteer satisfaction | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Brian D. Raffety, PhD, Principal Investigator — The Circumplex Company
Locations (1):
- The Circumplex Company, Seattle, Washington, United States